CLINICAL TRIAL: NCT02278276
Title: A Randomised, Double-blinded, Placebo-controlled Study to Assess the Safety and Bioactivity of Sodium Polysulthionate (SG1002) in Heart Failure Patients
Brief Title: Assessing the Safety and Bioactivity of SG1002 in Heart Failure Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sulfagenix Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sulfagenix-SG1002-002
Record Dates: First submitted 2014-10-23; First posted 2014-10-29 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0 mg SG1002 (Placebo Comparator): Capsules containing 400 mg of placebo will be provided to subjects. Subjects will take two tablets twice each day.
  Interventions: Drug: Placebo
- 1600 mg SG1002 (Active Comparator): Capsules containing 400 mg of sodium polysulthionate (SG1002) will be provided to subjects. Subjects will take two tablets twice each day, providing subjects with 1600 mg SG1002 daily.
  Interventions: Drug: sodium polysulthionate

INTERVENTIONS:
Drug: sodium polysulthionate — Bioavailable composition of α-sulfur
  Arms: 1600 mg SG1002
Drug: Placebo — 400 mg capsules containing placebo
  Arms: 0 mg SG1002

SUMMARY:
The purpose of this study is to determine the safety and benefits of SG1002, including overcoming deficits in circulating hydrogen sulfide and nitrite found in heart failure patients, with secondary endpoints focused on improving clinical endpoints.

DETAILED DESCRIPTION:
This will be a 3 month, placebo controlled double blind study, to determine whether 800 mg SG1002 given twice daily will be safe and will improve circulating levels of hydrogen sulfide and/or nitrite in heart failure subjects. In addition, secondary endpoints such as 6 minute walk distance, Minnesota heart failure questionnaire, biomarkers of inflammation and oxidative stress and cardiac remodeling will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic heart failure, with New York Heart Association (NYHA) classification of stage III;
* be ambulatory;
* have left ventricular ejection fraction less than 40% within 6 months of screening;
* have heart failure that has been stable for the previous 3 months (defined by no change in baseline therapy or symptoms of heart failure for the previous 3 months)(changes in diuretics are permitted);
* if female, be either post-menopausal or surgically sterilised or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) from signing of the informed consent form though to the Final Visit/Early Termination Visit; and
* be willing and able to provide written informed consent.

Exclusion Criteria:

* pregnant or breastfeeding;
* has had any of the following within 3 months prior to screening: myocardial infarction, unstable angina, cerebrovascular accident, percutaneous coronary intervention, open heart surgery, cardiac resynchronisation therapy (CRT) or transient ischaemic attack (TIA);
* has serious cerebrovascular disease in the opinion of the PI;
* is unable to walk without the assistance of another person;
* has primary lung disease that is the major contributor to current symptom status;
* is currently participating in another interventional clinical study, or has participated in one within 30 days prior to screening;
* has an inability to speak English (due to need to administer standardised English-language questionnaires);
* has current symptomatic hypotension (defined as systolic blood pressure (SBP) ≤ 90 mmHg or diastolic blood pressure (DBP) ≤ 40 mmHg);
* has poorly controlled hypertension (defined as SBP ≥ 160 mmHg or DBP ≥ 100 mmHg) despite therapy;
* will have percutaneous coronary intervention or open heart surgery within 3 months of the screening visit;
* has serious liver disease;
* has poorly controlled diabetes (defined as HbA1c > 10.0 %);
* has hypersensitivity to sulfur or related compounds;
* uses sulfur containing products or supplements, such as dimethyl sulfoxide (DMSO) or methylsulfonylmethane (MSM);
* has renal insufficiency defined as eGFR < 30 mL/minute/1.73 m2 (Modification of Diet in Renal Disease Study MDRD);
* has a life expectancy of less than 6 months;
* has active malignancy requiring active anti-neoplastic therapy that will, in the opinion of the Investigator, interfere with study treatment or participation. (Stable basal cell skin cancer and cancers being treated solely with hormonal therapy are allowed);
* has evidence of drug or alcohol abuse within the past 3 years;
* has any other chronic illness that may, in the opinion of the Investigator, increase the risks associated with this trial.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Composite measure using adverse events, clinical laboratory tests, vital signs and ECGs | 3 month
Changes in blood levels of hydrogen sulfide and nitrite in the SG1002 group measured by comparing the area under the curves after administration of the first dose and baseline levels of each at the first visit versus the final visit. | 3 months
  Demonstration of bioactivity as evidenced by increases in circulating levels of hydrogen sulfide and/or one or more nitric oxide metabolites, including nitrite, S-nitrosothiols and guanosine cyclic monophosphate levels as assessed by comparing AUC between placebo and SG1002 groups and by comparing baseline levels pre-administration at the start of the study to preadministration at the conclusion of the study.

SECONDARY OUTCOMES:
Heart function | 3 months
  A change from baseline to 13 weeks in BNP levels or cardiac remodeling as assessed by echocardiograms
Body mass and waste circumference | 3 months
  A change from baseline to 13 weeks in waist circumference and body mass index
Biomarkers of inflammation and oxidative stress | 3 months
  A change from baseline to 13 weeks in biomarkers of inflammation, C-reactive Protein (CRP) and interleukin 6 (IL6) and oxidative stress, oxidized LDL (oxLDL) and ratio of reduced glytathione (GSH) to oxidized glutathione (GSSG)
Walking distance in 6 minute | 3 months
  A change from baseline to 13 weeks in the distance walked in 6 minutes
Minnesota Heart Failure Questionnaire | 3 months
  A change from baseline to 13 weeks in quality of life as assessed by Minnesota Heart Failure Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tony Giordano, PhD, Study Director — Sulfagenix Australia Pty Ltd.